CLINICAL TRIAL: NCT05814640
Title: Sequenced Treatment Alternatives to Relieve Adolescent Depression (STAR-AD): a Pragmatic Clinical Trial
Brief Title: Sequenced Treatment Alternatives to Relieve Adolescent Depression (STAR-AD)
Acronym: STAR-AD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Second Xiangya Hospital of Central South University (Other); Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1stChongqingMU--ZXY
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depression; Sequestra
MeSH Terms: conditions — Depression | interventions — Fluoxetine; Sertraline; Vortioxetine; Duloxetine Hydrochloride; Aripiprazole; Lithium Carbonate; Olanzapine

STUDY DESIGN:
Intervention Model Description: After receiving fluoxetine and fluoxetine combined with cognitive-behavioral therapy, the next stage of treatment is determined by the patient's response (remission and non-remission) and is scheduled according to the patient's wishes and random assignment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the patient and the psychiatrist know which group they are allocated to, while the outcome assessor and data analyst are kept blind to the allocation. The clinicians providing the intervention do not perform the assessment and are unaware of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Fluoxetine (Experimental): Dosage form: po Dosage: 10-60mg Frequency: qn Course of treatment: 8 weeks. At week 8, patients will be evaluated as "in " or "not in remission." "Patients who are not in remission" will be randomized to phase II treatment based on the patient's wishes.
  Interventions: Drug: Fluoxetine
- group cognitive behavioral therapy（GCBT） (Experimental): GCBT was administered in addition to fluoxetine and consisted of 11 sessions for 8 weeks. It lasts 90 to 120 minutes, once or twice a week. At week 8, patients will be evaluated as "in remission" or "not in remission." "Patients who are not in remission" will be randomized to phase II treatment based on the patient's wishes.
  Interventions: Behavioral: GCBT
- Sertraline (Experimental): dosage form: po dosage:25-200mg frequency:qn duration: At Week 8, patients assessed as 'non-remission' will be given Sertraline as a switching treatment to fluoxetine.
  Interventions: Drug: Sertraline
- Vortioxetine (Experimental): dosage form: po dosage: 10-20mg frequency:qn duration: At Week 8, patients assessed as 'non-remission' will be given votioxetine as a switching treatment to fluoxetine.
  Interventions: Drug: Vortioxetine
- Duloxetine (Experimental): dosage form: po dosage: 60-120mg frequency: qn duration: At Week 8, patients assessed as 'non-remission' will be given duloxetine as an add-on treatment to fluoxetine.
  Interventions: Drug: Duloxetine
- Aripiprazole (Experimental): dosage form: po dosage: 2.5-15mg frequency:qn duration: At Week 8, patients assessed as 'non-remission' will be given aripiprazole as an add-on treatment to fluoxetine.
  Interventions: Drug: Aripiprazole
- Lithium carbonate (Experimental): dosage form: po dosage: 125-500mg frequency: qn duration: At Week 8, patients assessed as 'non-response' will be given lithium carbonate as an add-on treatment to fluoxetine.
  Interventions: Drug: Lithium Carbonate
- Olanzapine (Experimental): dosage form:po dosage: 1.25-10mg frequency:qn duration: At Week 8, patients assessed as 'non-rremission' will be given olanzapine as an add-on treatment to fluoxetine.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Fluoxetine — Commonly used oral antidepressant.
  Arms: Fluoxetine
Drug: Sertraline — Commonly used oral antidepressant.
  Arms: Sertraline
Drug: Vortioxetine — Commonly used oral antidepressant.
  Arms: Vortioxetine
Drug: Duloxetine — Commonly used oral antidepressant.
  Arms: Duloxetine
Drug: Aripiprazole — Commonly used oral augmentation therapy for antidepressants
  Arms: Aripiprazole
Drug: Lithium Carbonate — Commonly used oral augmentation therapy for antidepressants.
  Arms: Lithium carbonate
Drug: Olanzapine — Commonly used oral augmentation therapy for antidepressants.
  Arms: Olanzapine
Behavioral: GCBT — Commonly used intervention therapy of psychotherapy.
  Arms: group cognitive behavioral therapy（GCBT）

SUMMARY:
This project aims to investigate the effectiveness of existing common antidepressants and to provide new evidence for depressed children and adolescents who are not responding to their first treatment.

DETAILED DESCRIPTION:
This is an open-label Sequential Multiple Assignment Randomized Trial (SMART) of 16 weeks duration with two levels, each stage 8 weeks. In phase 1, adolescents with MDD will be selected into fluoxetine or fluoxetine combination CBT therapy groups and the choice of treatment will be at the discretion of the patient. Subjects who fail to respond will enter phase 2 randomization， where patients will be randomly assigned to oral sertraline, votioxetine, duloxetine or adding one of aripiprazole, lithium carbonate, and olanzapine to fluoxetine. The primary outcome of the treatment phase is the treatment remission rate and response rate. Secondary outcomes included: symptom scale; Quality of life; Sleep therapy; Symptoms of anxiety; Rumination and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13 - 18
2. As assessed by K-SADS-PL, it meets the DSM-V criteria for MDD with non-psychotic symptoms
3. Score≥40 on the CDRS-R
4. Participants with suicidal ideation are eligible, as long as clinicians consider outpatient treatment to be safe
5. Sufficient audio-visual level to complete this study
6. Written informed consent was obtained from patients and at least one of their parents

Exclusion Criteria:

1. History of bipolar disorder, schizophrenia, autism, eating disorders, primary obsessive compulsive disorder, pervasive developmental disorder, or psychosis not otherwise specified
2. History of serious physical illnesses
3. Substance abuse or dependence
4. Current depressive episode with clear suicidal plans or suicidal behavior
5. Requires inpatient treatment for psychiatric disorders
6. Severe mental disorders requiring
7. 2 or more failed trials of antidepressant drugs: each trial for at least 8 weeks, with the last 4 weeks at full dose (e.g. fluoxetine 40mg/d, citalopram 40mg/d, escitalopram 20mg/d, sertraline 150mg/d )
8. History of clear-cut intolerability of, or lack of effect with, an adequate trial of at least one protocol treatment option
9. Taking any medicine that contraindicates in combination with or interferes with the efficacy of the treatment
10. Taking or administering antidepressants within 5 half-lives
11. Received modified electroconvulsive therapy within 12 months
12. If female, is pregnant

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in CDRS-R (Children's Depression Rating Scale) scores from baseline | Baseline of treatment period, 2 weeks, 1 month, 2 months, 3 months，4months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  Clinical response (≥ 50% reduction in CDRS-R scores from baseline)

SECONDARY OUTCOMES:
Change in BDI-II (Baker Depression Scale) scores from baseline | Baseline of treatment period, 1 month, 2 months, 3 months，4 months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  Change in BDI-II (Baker Depression Scale) scores from baseline
Change in SCARED (The Screen for Child Anxiety-Related Emotional Disorders) scores from baseline | Baseline of treatment period, 1 month, 2 months, 3 months，4 months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  Improvement in anxiety (SCARED minus the scores）
Change in suicide risk from baseline on the C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline of treatment period, 1 month, 2 months, 3 months，4 months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  The severity of the suicide risk
Change in PSQI (Pittsburgh Sleep Quality Index) scores from baseline | Baseline of treatment period, 2 month, 4 months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  Improvement in sleep status (PSQI minus the scores）
Change in PedsQL4.0 (The Pediatric Quality of Life Inventory) scores from baseline | Baseline of treatment period, 2 month, 4 months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  Improvement of children's quality of life（PedsQL4.0 minus the scores)
Change in CGI-S (Clinical Global Impressions-Severity Scales) scores from baseline | Baseline of treatment period, 1 month, 2 months, 3 months，4 months.
  Improvement in overall clinical impression severity（ 7-point scale, with 1 being normal and 7 being among the most severely damaged）
Change in CGI-I (Clinical Global Impressions-Improvement Scales) scores from baseline | The treatment period was 1 month, 2 months, 3 months，4 months.
  Improvement of clinical general Impression scale（ 7-point scale,7 denoting a very significant deterioration）
Change in RSS (Ruminative Responses Scale) | The treatment period was 1 month, 2 months.
  The level of improvement in negative thinking（he higher the total score, the more reflective thinking The more severe it is）
Change in HCL-32（Hypomania Symptom Checklist-32） | Baseline of treatment period, 1 month, 2 months, 3 months，4 months; The follow-up period was 1 month, 3 months, 6 months and 12 months
  Assess the patient's hypomanic state

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Province, China

REFERENCES:
- [Background] Gunlicks-Stoessel M, Mufson L, Bernstein G, Westervelt A, Reigstad K, Klimes-Dougan B, Cullen K, Murray A, Vock D. Critical Decision Points for Augmenting Interpersonal Psychotherapy for Depressed Adolescents: A Pilot Sequential Multiple Assignment Randomized Trial. J Am Acad Child Adolesc Psychiatry. 2019 Jan;58(1):80-91. doi: 10.1016/j.jaac.2018.06.032. Epub 2018 Oct 27. PMID 30577943
- [Background] Hawton K, van Heeringen K. Suicide. Lancet. 2009 Apr 18;373(9672):1372-81. doi: 10.1016/S0140-6736(09)60372-X. PMID 19376453
- [Background] van Ettekoven KM, Rasing SPA, Vermulst AA, Engels RCME, Kindt KCM, Creemers DHM. Cross-Lagged Associations between Depressive Symptoms and Response Style in Adolescents. Int J Environ Res Public Health. 2020 Feb 21;17(4):1380. doi: 10.3390/ijerph17041380. PMID 32098035
- [Background] Twenge JM, Cooper AB, Joiner TE, Duffy ME, Binau SG. Age, period, and cohort trends in mood disorder indicators and suicide-related outcomes in a nationally representative dataset, 2005-2017. J Abnorm Psychol. 2019 Apr;128(3):185-199. doi: 10.1037/abn0000410. Epub 2019 Mar 14. PMID 30869927
- [Background] McCarty CA, Weisz JR. Effects of psychotherapy for depression in children and adolescents: what we can (and can't) learn from meta-analysis and component profiling. J Am Acad Child Adolesc Psychiatry. 2007 Jul;46(7):879-86. doi: 10.1097/chi.0b013e31805467b3. PMID 17581452
- [Background] Birmaher B, Brent D; AACAP Work Group on Quality Issues; Bernet W, Bukstein O, Walter H, Benson RS, Chrisman A, Farchione T, Greenhill L, Hamilton J, Keable H, Kinlan J, Schoettle U, Stock S, Ptakowski KK, Medicus J. Practice parameter for the assessment and treatment of children and adolescents with depressive disorders. J Am Acad Child Adolesc Psychiatry. 2007 Nov;46(11):1503-26. doi: 10.1097/chi.0b013e318145ae1c. PMID 18049300
- [Background] Luxton R, Kyriakopoulos M. Depression in children and young people: identification and management NICE guidelines. Arch Dis Child Educ Pract Ed. 2022 Feb;107(1):36-38. doi: 10.1136/archdischild-2020-320020. Epub 2021 May 10. No abstract available. PMID 33972346
- [Background] MacQueen GM, Frey BN, Ismail Z, Jaworska N, Steiner M, Lieshout RJ, Kennedy SH, Lam RW, Milev RV, Parikh SV, Ravindran AV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 6. Special Populations: Youth, Women, and the Elderly. Can J Psychiatry. 2016 Sep;61(9):588-603. doi: 10.1177/0706743716659276. Epub 2016 Aug 2. PMID 27486149
- [Background] Cheung AH, Zuckerbrot RA, Jensen PS, Laraque D, Stein REK; GLAD-PC STEERING GROUP. Guidelines for Adolescent Depression in Primary Care (GLAD-PC): Part II. Treatment and Ongoing Management. Pediatrics. 2018 Mar;141(3):e20174082. doi: 10.1542/peds.2017-4082. PMID 29483201
- [Background] Feng Y, Xiao L, Wang WW, Ungvari GS, Ng CH, Wang G, Xiang YT. Guidelines for the diagnosis and treatment of depressive disorders in China: The second edition. J Affect Disord. 2019 Jun 15;253:352-356. doi: 10.1016/j.jad.2019.04.104. Epub 2019 May 1. PMID 31078835
- [Background] March J, Silva S, Petrycki S, Curry J, Wells K, Fairbank J, Burns B, Domino M, McNulty S, Vitiello B, Severe J; Treatment for Adolescents With Depression Study (TADS) Team. Fluoxetine, cognitive-behavioral therapy, and their combination for adolescents with depression: Treatment for Adolescents With Depression Study (TADS) randomized controlled trial. JAMA. 2004 Aug 18;292(7):807-20. doi: 10.1001/jama.292.7.807. PMID 15315995
- [Background] Mufson L, Dorta KP, Wickramaratne P, Nomura Y, Olfson M, Weissman MM. A randomized effectiveness trial of interpersonal psychotherapy for depressed adolescents. Arch Gen Psychiatry. 2004 Jun;61(6):577-84. doi: 10.1001/archpsyc.61.6.577. PMID 15184237
- [Background] Brent D, Emslie G, Clarke G, Wagner KD, Asarnow JR, Keller M, Vitiello B, Ritz L, Iyengar S, Abebe K, Birmaher B, Ryan N, Kennard B, Hughes C, DeBar L, McCracken J, Strober M, Suddath R, Spirito A, Leonard H, Melhem N, Porta G, Onorato M, Zelazny J. Switching to another SSRI or to venlafaxine with or without cognitive behavioral therapy for adolescents with SSRI-resistant depression: the TORDIA randomized controlled trial. JAMA. 2008 Feb 27;299(8):901-913. doi: 10.1001/jama.299.8.901. PMID 18314433
- [Background] Emslie GJ, Mayes T, Porta G, Vitiello B, Clarke G, Wagner KD, Asarnow JR, Spirito A, Birmaher B, Ryan N, Kennard B, DeBar L, McCracken J, Strober M, Onorato M, Zelazny J, Keller M, Iyengar S, Brent D. Treatment of Resistant Depression in Adolescents (TORDIA): week 24 outcomes. Am J Psychiatry. 2010 Jul;167(7):782-91. doi: 10.1176/appi.ajp.2010.09040552. Epub 2010 May 17. PMID 20478877
- [Background] El-Hage W. [Roadmap for therapeutic strategies of treatment resistant depression]. Presse Med. 2016 Mar;45(3):320-2. doi: 10.1016/j.lpm.2016.02.001. Epub 2016 Mar 9. No abstract available. French. PMID 26970939
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Background] Sinyor M, Schaffer A, Levitt A. The sequenced treatment alternatives to relieve depression (STAR*D) trial: a review. Can J Psychiatry. 2010 Mar;55(3):126-35. doi: 10.1177/070674371005500303. PMID 20370962
- [Background] Trivedi MH, Fava M, Wisniewski SR, Thase ME, Quitkin F, Warden D, Ritz L, Nierenberg AA, Lebowitz BD, Biggs MM, Luther JF, Shores-Wilson K, Rush AJ; STAR*D Study Team. Medication augmentation after the failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1243-52. doi: 10.1056/NEJMoa052964. PMID 16554526
- [Background] Malhi GS, Bassett D, Boyce P, Bryant R, Fitzgerald PB, Fritz K, Hopwood M, Lyndon B, Mulder R, Murray G, Porter R, Singh AB. Royal Australian and New Zealand College of Psychiatrists clinical practice guidelines for mood disorders. Aust N Z J Psychiatry. 2015 Dec;49(12):1087-206. doi: 10.1177/0004867415617657. PMID 26643054
- [Background] Cleare A, Pariante CM, Young AH, Anderson IM, Christmas D, Cowen PJ, Dickens C, Ferrier IN, Geddes J, Gilbody S, Haddad PM, Katona C, Lewis G, Malizia A, McAllister-Williams RH, Ramchandani P, Scott J, Taylor D, Uher R; Members of the Consensus Meeting. Evidence-based guidelines for treating depressive disorders with antidepressants: A revision of the 2008 British Association for Psychopharmacology guidelines. J Psychopharmacol. 2015 May;29(5):459-525. doi: 10.1177/0269881115581093. Epub 2015 May 12. PMID 25969470
- [Background] Bauer M, Pfennig A, Severus E, Whybrow PC, Angst J, Moller HJ; World Federation of Societies of Biological Psychiatry. Task Force on Unipolar Depressive Disorders. World Federation of Societies of Biological Psychiatry (WFSBP) guidelines for biological treatment of unipolar depressive disorders, part 1: update 2013 on the acute and continuation treatment of unipolar depressive disorders. World J Biol Psychiatry. 2013 Jul;14(5):334-85. doi: 10.3109/15622975.2013.804195. Epub 2013 Jul 3. PMID 23879318
- [Background] DeBattista C, Doghramji K, Menza MA, Rosenthal MH, Fieve RR; Modafinil in Depression Study Group. Adjunct modafinil for the short-term treatment of fatigue and sleepiness in patients with major depressive disorder: a preliminary double-blind, placebo-controlled study. J Clin Psychiatry. 2003 Sep;64(9):1057-64. doi: 10.4088/jcp.v64n0911. PMID 14628981
- [Background] Murphy SA. An experimental design for the development of adaptive treatment strategies. Stat Med. 2005 May 30;24(10):1455-81. doi: 10.1002/sim.2022. PMID 15586395
- [Background] Ogbagaber SB, Karp J, Wahed AS. Design of sequentially randomized trials for testing adaptive treatment strategies. Stat Med. 2016 Mar 15;35(6):840-58. doi: 10.1002/sim.6747. Epub 2015 Sep 27. PMID 26412033
- [Background] Liu Y, Zeng D, Wang Y. Use of personalized Dynamic Treatment Regimes (DTRs) and Sequential Multiple Assignment Randomized Trials (SMARTs) in mental health studies. Shanghai Arch Psychiatry. 2014 Dec;26(6):376-83. doi: 10.11919/j.issn.1002-0829.214172. PMID 25642116
- [Background] Frank E, Prien RF, Jarrett RB, Keller MB, Kupfer DJ, Lavori PW, Rush AJ, Weissman MM. Conceptualization and rationale for consensus definitions of terms in major depressive disorder. Remission, recovery, relapse, and recurrence. Arch Gen Psychiatry. 1991 Sep;48(9):851-5. doi: 10.1001/archpsyc.1991.01810330075011. PMID 1929776
- [Background] Cheung A, Kusumakar V, Kutcher S, Dubo E, Garland J, Weiss M, Kiss A, Levitt A. Maintenance study for adolescent depression. J Child Adolesc Psychopharmacol. 2008 Aug;18(4):389-94. doi: 10.1089/cap.2008.0001. PMID 18759650
- [Background] Emslie GJ, Mayes TL. Mood disorders in children and adolescents: psychopharmacological treatment. Biol Psychiatry. 2001 Jun 15;49(12):1082-90. doi: 10.1016/s0006-3223(01)01149-0. PMID 11430850
- [Background] Emslie GJ, Heiligenstein JH, Wagner KD, Hoog SL, Ernest DE, Brown E, Nilsson M, Jacobson JG. Fluoxetine for acute treatment of depression in children and adolescents: a placebo-controlled, randomized clinical trial. J Am Acad Child Adolesc Psychiatry. 2002 Oct;41(10):1205-15. doi: 10.1097/00004583-200210000-00010. PMID 12364842
- [Background] Thome-Souza MS, Kuczynski E, Valente KD. Sertraline and fluoxetine: safe treatments for children and adolescents with epilepsy and depression. Epilepsy Behav. 2007 May;10(3):417-25. doi: 10.1016/j.yebeh.2007.01.004. Epub 2007 Feb 15. PMID 17306625
- [Background] Zhou X, Teng T, Zhang Y, Del Giovane C, Furukawa TA, Weisz JR, Li X, Cuijpers P, Coghill D, Xiang Y, Hetrick SE, Leucht S, Qin M, Barth J, Ravindran AV, Yang L, Curry J, Fan L, Silva SG, Cipriani A, Xie P. Comparative efficacy and acceptability of antidepressants, psychotherapies, and their combination for acute treatment of children and adolescents with depressive disorder: a systematic review and network meta-analysis. Lancet Psychiatry. 2020 Jul;7(7):581-601. doi: 10.1016/S2215-0366(20)30137-1. PMID 32563306
- [Background] Wagner KD, Ambrosini P, Rynn M, Wohlberg C, Yang R, Greenbaum MS, Childress A, Donnelly C, Deas D; Sertraline Pediatric Depression Study Group. Efficacy of sertraline in the treatment of children and adolescents with major depressive disorder: two randomized controlled trials. JAMA. 2003 Aug 27;290(8):1033-41. doi: 10.1001/jama.290.8.1033. PMID 12941675
- [Background] Cipriani A, Zhou X, Del Giovane C, Hetrick SE, Qin B, Whittington C, Coghill D, Zhang Y, Hazell P, Leucht S, Cuijpers P, Pu J, Cohen D, Ravindran AV, Liu Y, Michael KD, Yang L, Liu L, Xie P. Comparative efficacy and tolerability of antidepressants for major depressive disorder in children and adolescents: a network meta-analysis. Lancet. 2016 Aug 27;388(10047):881-90. doi: 10.1016/S0140-6736(16)30385-3. Epub 2016 Jun 8. PMID 27289172
- [Background] Hetrick SE, McKenzie JE, Bailey AP, Sharma V, Moller CI, Badcock PB, Cox GR, Merry SN, Meader N. New generation antidepressants for depression in children and adolescents: a network meta-analysis. Cochrane Database Syst Rev. 2021 May 24;5(5):CD013674. doi: 10.1002/14651858.CD013674.pub2. PMID 34029378
- [Background] Bang-Andersen B, Ruhland T, Jorgensen M, Smith G, Frederiksen K, Jensen KG, Zhong H, Nielsen SM, Hogg S, Mork A, Stensbol TB. Discovery of 1-[2-(2,4-dimethylphenylsulfanyl)phenyl]piperazine (Lu AA21004): a novel multimodal compound for the treatment of major depressive disorder. J Med Chem. 2011 May 12;54(9):3206-21. doi: 10.1021/jm101459g. Epub 2011 Apr 12. PMID 21486038
- [Background] Findling RL, DelBello MP, Zuddas A, Emslie GJ, Ettrup A, Petersen ML, Schmidt SN, Rosen M. Vortioxetine for Major Depressive Disorder in Adolescents: 12-Week Randomized, Placebo-Controlled, Fluoxetine-Referenced, Fixed-Dose Study. J Am Acad Child Adolesc Psychiatry. 2022 Sep;61(9):1106-1118.e2. doi: 10.1016/j.jaac.2022.01.004. Epub 2022 Jan 13. PMID 35033635
- [Background] Makrogiannis S, Zheng K, Harris C. Discriminative Localized Sparse Approximations for Mass Characterization in Mammograms. Front Oncol. 2021 Dec 30;11:725320. doi: 10.3389/fonc.2021.725320. eCollection 2021. PMID 35036353
- [Background] Thase ME, Mahableshwarkar AR, Dragheim M, Loft H, Vieta E. A meta-analysis of randomized, placebo-controlled trials of vortioxetine for the treatment of major depressive disorder in adults. Eur Neuropsychopharmacol. 2016 Jun;26(6):979-93. doi: 10.1016/j.euroneuro.2016.03.007. Epub 2016 Mar 25. PMID 27139079
- [Background] Cipriani A, Furukawa TA, Salanti G, Chaimani A, Atkinson LZ, Ogawa Y, Leucht S, Ruhe HG, Turner EH, Higgins JPT, Egger M, Takeshima N, Hayasaka Y, Imai H, Shinohara K, Tajika A, Ioannidis JPA, Geddes JR. Comparative efficacy and acceptability of 21 antidepressant drugs for the acute treatment of adults with major depressive disorder: a systematic review and network meta-analysis. Lancet. 2018 Apr 7;391(10128):1357-1366. doi: 10.1016/S0140-6736(17)32802-7. Epub 2018 Feb 21. PMID 29477251
- [Background] Nunez NA, Joseph B, Pahwa M, Kumar R, Resendez MG, Prokop LJ, Veldic M, Seshadri A, Biernacka JM, Frye MA, Wang Z, Singh B. Augmentation strategies for treatment resistant major depression: A systematic review and network meta-analysis. J Affect Disord. 2022 Apr 1;302:385-400. doi: 10.1016/j.jad.2021.12.134. Epub 2022 Jan 2. PMID 34986373
- [Background] Seshadri A, Wermers ME, Habermann TJ, Singh B. Long-term Efficacy and Tolerability of Adjunctive Aripiprazole for Major Depressive Disorder: Systematic Review and Meta-analysis. Prim Care Companion CNS Disord. 2021 Jun 24;23(4):20r02799. doi: 10.4088/PCC.20r02799. PMID 34167174
- [Background] Strawbridge R, Carter B, Marwood L, Bandelow B, Tsapekos D, Nikolova VL, Taylor R, Mantingh T, de Angel V, Patrick F, Cleare AJ, Young AH. Augmentation therapies for treatment-resistant depression: systematic review and meta-analysis. Br J Psychiatry. 2019 Jan;214(1):42-51. doi: 10.1192/bjp.2018.233. Epub 2018 Nov 20. PMID 30457075
- [Background] Kennedy SH, Lam RW, McIntyre RS, Tourjman SV, Bhat V, Blier P, Hasnain M, Jollant F, Levitt AJ, MacQueen GM, McInerney SJ, McIntosh D, Milev RV, Muller DJ, Parikh SV, Pearson NL, Ravindran AV, Uher R; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 3. Pharmacological Treatments. Can J Psychiatry. 2016 Sep;61(9):540-60. doi: 10.1177/0706743716659417. Epub 2016 Aug 2. PMID 27486148
- [Background] Spielmans GI, Berman MI, Linardatos E, Rosenlicht NZ, Perry A, Tsai AC. Adjunctive Atypical Antipsychotic Treatment for Major Depressive Disorder: A Meta-Analysis of Depression, Quality of Life, and Safety Outcomes. Focus (Am Psychiatr Publ). 2016 Apr;14(2):244-265. doi: 10.1176/appi.focus.140202. Epub 2016 Apr 7. PMID 31997952
- [Background] Vazquez GH, Bahji A, Undurraga J, Tondo L, Baldessarini RJ. Efficacy and Tolerability of Combination Treatments for Major Depression: Antidepressants plus Second-Generation Antipsychotics vs. Esketamine vs. Lithium. J Psychopharmacol. 2021 Aug;35(8):890-900. doi: 10.1177/02698811211013579. Epub 2021 Jul 9. PMID 34238049
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430
- [Background] Su L, Wang K, Fan F, Su Y, Gao X. Reliability and validity of the screen for child anxiety related emotional disorders (SCARED) in Chinese children. J Anxiety Disord. 2008 May;22(4):612-21. doi: 10.1016/j.janxdis.2007.05.011. Epub 2007 Jun 3. PMID 17628391
- [Background] Phillips MR, Li X, Zhang Y. Suicide rates in China, 1995-99. Lancet. 2002 Mar 9;359(9309):835-40. doi: 10.1016/S0140-6736(02)07954-0. PMID 11897283
- [Background] Viguera AC, Milano N, Laurel R, Thompson NR, Griffith SD, Baldessarini RJ, Katzan IL. Comparison of Electronic Screening for Suicidal Risk With the Patient Health Questionnaire Item 9 and the Columbia Suicide Severity Rating Scale in an Outpatient Psychiatric Clinic. Psychosomatics. 2015 Sep-Oct;56(5):460-9. doi: 10.1016/j.psym.2015.04.005. Epub 2015 May 8. PMID 26278339
- [Background] Angst J, Adolfsson R, Benazzi F, Gamma A, Hantouche E, Meyer TD, Skeppar P, Vieta E, Scott J. The HCL-32: towards a self-assessment tool for hypomanic symptoms in outpatients. J Affect Disord. 2005 Oct;88(2):217-33. doi: 10.1016/j.jad.2005.05.011. PMID 16125784
- [Background] Yang HC, Yuan CM, Liu TB, Li LJ, Peng HJ, Liao CP, Rong H, Fang YR, Angst J. Validity of the 32-item Hypomania Checklist (HCL-32) in a clinical sample with mood disorders in China. BMC Psychiatry. 2011 May 15;11:84. doi: 10.1186/1471-244X-11-84. PMID 21575151
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Nolen-Hoeksema S, Morrow J. A prospective study of depression and posttraumatic stress symptoms after a natural disaster: the 1989 Loma Prieta Earthquake. J Pers Soc Psychol. 1991 Jul;61(1):115-21. doi: 10.1037//0022-3514.61.1.115. PMID 1890582
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Li TJ, Sun YC, Ma QY, Wu Y, Yang C, Zhang N, Yang Y, Yang YX. Clinical observation of Dan-Hong Hua-Yu oral solution in treating retinal vein occlusion. Medicine (Baltimore). 2020 May 22;99(21):e20173. doi: 10.1097/MD.0000000000020173. PMID 32481287
- [Derived] He Y, Gan X, Li X, Wang T, Li J, Lei T, Huang Y, Liu R, Chen F, Teng T, Xie Y, Ouyang X, Zhou X. Sequenced treatment alternatives to relieve adolescent depression (STAR-AD): a multicentre open-label randomized controlled trial protocol. BMC Psychiatry. 2023 Oct 27;23(1):789. doi: 10.1186/s12888-023-05221-w. PMID 37891522
- See also: Depression and Other Common Mental Disorders Global Health Estimates — http://apps.who.int/iris/handle/10665/254610
- See also: Depression in adults: recognition and management — https://www.nice.org.uk/guidance/ng222
- See also: Review and opportunity analysis of antidepressant drug market in China — https://www.menet.com.cn/